CLINICAL TRIAL: NCT04838613
Title: Phase III Study for Evaluation of the Diagnostic Performance of [18F]CTT1057 PET Imaging in Patients With Prostate Cancer With Rising PSA Levels [Biochemical Recurrence (BCR)]
Brief Title: Study of Diagnostic Performance of [18F]CTT1057 in BCR
Acronym: GuidePath
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAA405A12301; 2020-003959-16 (EudraCT Number)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Prostatic Neoplasms; Prostate Cancer; Recurrence
Keywords: [18F]CTT1057; [68Ga]Ga-PSMA-11; Positron Emission Tomography/Computerized Tomography; PET/CT; Radioligand; Imaging; Biochemical recurrence; BCR; Composite Truth Standard; CTS; Prostate Cancer; PCa
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: Once eligibility was confirmed, the participants were randomized in IRT to be assigned to one of the following two PET/CT scan sequences at random in a 1:1 ratio:
  * Sequence 1: [18F]CTT1057 on Day 1 (investigational imaging agent of interest) followed by [68Ga]Ga-PSMA-11 at least 14 days apart (as part of CTS if required, and for secondary endpoint)
  * Sequence 2: [68Ga]Ga-PSMA-11 (as part of CTS if required, and for secondary endpoint) on Day 1 followed by [18F]CTT1057 (investigational imaging agent of interest) at least 14 days apart
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET/CT imaging with [18F]CTT1057 followed by [68Ga]Ga-PSMA-11 or vice versa (Experimental): All eligible participants were assigned to one of the following two PET/CT scan sequences at random in a 1:1 ratio:
  * Sequence 1: [18F]CTT1057 on Day 1 (investigational imaging agent of interest) followed by [68Ga]Ga-PSMA-11 at least 14 days apart (as part of CTS if required, and for secondary endpoint)
  * Sequence 2: [68Ga]Ga-PSMA-11 (as part of CTS if required, and for secondary endpoint) on Day 1 followed by [18F]CTT1057 (investigational imaging agent of interest) at least 14 days apart
  Interventions: Drug: [18F]CTT1057; Drug: [68Ga]Ga-PSMA-11

INTERVENTIONS:
Drug: [18F]CTT1057 — Single intravenous dose of approximately 370 Mega-Becquerel (MBq) and subsequent PET/CT scan
Drug: [68Ga]Ga-PSMA-11 — Single intravenous dose of approximately 150 MBq and subsequent PET/CT scan

SUMMARY:
The current study aimed at evaluating the diagnostic performance of [18F]CTT1057 as a PET imaging agent for detection and localization of Prostate specific membrane antigen (PSMA) positivity in patients diagnosed of biochemical recurrence of prostate cancer (PCa), using a composite truth standard.

Approximately 190 participants were to be enrolled to ensure at least 152 participants were evaluable (i.e. have both an evaluable [18F]CTT1057 Positron emission tomography/Computed Tomography (PET/CT) scan imaging and at least one evaluable Composite Truth Standard (CTS) assessment and had not received any prohibited systemic antineoplastic therapy before the completion of PET/CTs and CTS procedures, which were required for the calculation of the co-primary endpoints.

DETAILED DESCRIPTION:
This was a prospective, open-label, multi center, single-arm Phase III study to evaluate the diagnostic performance of [18F]CTT1057 as a PET imaging agent for detection and localization of PSMA positive tumors in PCa patients diagnosed with biochemical recurrence (BCR) after initial definitive therapy with either radical prostatectomy (RP) or curative intent radiation therapy (RT), using a CTS as reference.

The CTS to be used as reference were hierarchical in nature, with 3 levels of Standard of Truth (SoT) procedures, that were applied as follows:

CTS Level 1: Histopathology if available for the lesion (from prospective biopsy or salvage surgery performed within 8 weeks after the [18F]CTT1057 PET/CT scan); OR in case that histopathology was not available for a lesion, inconclusive or negative (for biopsy only).

CTS Level 2: Imaging diagnostic procedures performed on each patient as clinically indicated per SoC, which included at least a high resolution CT scan with contrast and a [68Ga]Ga-PSMA-11 PET/CT) performed within 8 weeks (either before or after) the [18F]CTT1057 PET/CT scan. Three-month follow-up imaging (from baseline) were also be used as part of the CTS level 2 in cases where it is clinically required for the diagnosis of particular lesion(s); OR if neither of the two above were feasible or deemed appropriate or they were inconclusive.

CTS Level 3: 50% or greater decline in PSA following radiation therapy (as long as no concomitant androgen deprivation therapy (ADT) was given) as per Prostate Cancer Working Group 3 (PCWG3) criteria.

All participants underwent 2 PET/CT scans: one with the investigational agent [18F]CTT1057 and another with [68Ga]Ga-PSMA-11 (as a component of the CTS Level 2 and for a secondary endpoint of assessment of concordance between the 2 PET/CT scans for detection of lesions). The 2 PET imaging procedures were performed at least 14 days apart, and the PET/CT scan sequence for each participant was assigned at random in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent must be obtained prior to participation in the study
* Biopsy proven prostate adenocarcinoma.
* Biochemical recurrence following initial definitive therapy (with either RP or curative intent radiation therapy) as defined:

by AUA criteria (Cookson et al 2007) for patients who have undergone RP: Initial serum PSA of ≥0.2 ng/ml measured at least 6 weeks after RP with a second confirmatory persistent PSA level of >0.2 ng/ml, or by ASTRO-Phoenix criteria (Roach et al 2006) for patients who have undergone curative-intent radiation therapy (RT): Rise of serum PSA measurement of 2 or more ng/mL above the nadir PSA observed post RT.

* ECOG performance status 0-2
* Participants must be adults ≥ 18 years of age

Exclusion Criteria:

* Inability to complete the needed investigational and standard-of-care imaging examinations due to any reason (severe claustrophobia, inability to lie still for the entire imaging time, etc.)
* Any additional medical condition, serious intercurrent illness, concomitant cancer or other extenuating circumstance that, in the opinion of the Investigator, would indicate a significant risk to safety or impair study participation, including, but not limited to, current severe urinary incontinence, hydronephrosis, severe voiding dysfunction, need of indwelling/condom catheters, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B or C, and COVID-19
* Prior major surgery undergone less than 12 weeks prior to screening (with the exception of any surgery related to prostatic cancer)
* Known allergy, hypersensitivity, or intolerance to [18F]CTT1057, [68Ga]Ga-PSMA-11, or to CT contrast
* Prior and current use of PSMA targeted therapies
* Prior ADT (first or second generation), including LHRH analogues (agonists or antagonists), within 9 months before screening
* Any 5-alpha reductase inhibitors within 30 days before screening
* Use of other investigational drugs within 30 days before screening
* Castration-resistant patients
* Patient with small cell or neuroendocrine PCa in more than 50% of biopsy tissue
* Prior salvage surgery or salvage radiation therapy

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Explorer Molecular Imaging center, Sacramento, California, United States
- France (5):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Toulouse
- Spain (4):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 190 participants were randomized using a 1:1 ratio to receive either Sequence 1 (vidoflufolastat (18F) followed by gallium (68Ga) gozetotide; N= 96) or Sequence 2 (gallium (68Ga) gozetotide followed by vidoflufolastat (18F); N=94). Out of the 190 randomized participants, 169 completed the study.
Pre-assignment Details: Prior to participation in the study, patients had to have biopsy proven prostate adenocarcinoma and diagnosis of biochemical recurrence following initial definitive therapy with either radical prostatectomy or curative intent radiation therapy.
Groups:
- PET/CT Imaging With Vidoflufolastat (18F) Followed by Gallium (68Ga) Gozetotide: Sequence 1: All eligible participants were assigned to this PET/CT scan sequence at random in a 1:1 ratio:
  - Sequence 1: vidoflufolastat (18F) on Day 1 (investigational imaging agent of interest) followed by gallium (68Ga) gozetotide at least 14 days apart (as part of CTS if required, and for secondary endpoint)
- PET/CT Imaging With Gallium (68Ga) Gozetotide Followed by Vidoflufolastat (18F): Sequence 2: All eligible participants were assigned to the following PET/CT scan sequence at random in a 1:1 ratio:
  - Sequence 2: gallium (68Ga) gozetotide (as part of CTS if required, and for secondary endpoint) on Day 1 followed by vidoflufolastat (18F) (investigational imaging agent of interest) at least 14 days apart
Period: Overall Study
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F) Followed by Gallium (68Ga) Gozetotide: Sequence 1 | PET/CT Imaging With Gallium (68Ga) Gozetotide Followed by Vidoflufolastat (18F): Sequence 2
Started | 96 | 94
Completed | 88 | 81
Not Completed | 8 | 13
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Protocol Deviation | 3 | 2
Not completed — Technical Problems | 0 | 5
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all randomized participants. Per protocol, two PET/CT scans were performed at least 2 weeks apart to ensure a clean safety profile assessment for each PET radiopharmaceutical. Participants were randomly assigned (1:1 ratio) to one of two scan sequences to counter-balance any potential change in lesions between the 2 scans:
  1. [18F]CTT1057 followed by [68Ga]Ga-PSMA-11
  2. [68Ga]Ga-PSMA-11 followed by [18F]CTT1057 Study was not intended to compare the two sequences.
Groups:
- PET/CT Imaging With Vidoflufolastat (18F) Followed by Gallium (68Ga) Gozetotide or Vice Versa: All eligible participants were assigned to one of the following two PET/CT scan sequences at random in a 1:1 ratio:- Sequence 1: vidoflufolastat (18F) on Day 1 (investigational imaging agent of interest) followed by gallium (68Ga) gozetotide at least 14 days apart (as part of CTS if required, and for secondary endpoint)- Sequence 2: gallium (68Ga) gozetotide (as part of CTS if required, and for secondary endpoint) on Day 1 followed by vidoflufolastat (18F) (investigational imaging agent of interest) at least 14 days apart
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F) Followed by Gallium (68Ga) Gozetotide or Vice Versa
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 180
  Black or African American | 4
  Asian | 2
  Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Region-level Correct Localization Rate (CLR) of Vidoflufolastat (18F)
Description: Region-level correct localization rate (CLR) is defined as the percentage of regions containing at least one True Positive (TP) lesion (exactly localized correspondence between PET imaging and the reference standard), regardless of any co-existent False Positive (FP) findings within the same region, out of all regions containing at least one PET-positive finding.
Time Frame: vidoflufolastat (18F) PET imaging acquired at Day 1 or Day 15 assessed against Composite Truth Standard (CTS) obtained within 8 weeks (before or after) of 18F-CTT PET scan or during follow-up (up to 90 days after radiotherapy for PSA level assessment)
Population: The Efficacy Analysis Set (EFF) included all randomized participants who received the dose of investigational treatment (i.e. vidoflufolastat (18F)), had both an evaluable vidoflufolastat (18F) PET/CT scan imaging and at least one evaluable CTS assessment, and did not receive any prohibited systemic antineoplastic therapy before the completion of PET/CTs and CTS procedures. Baseline PSA levels were unavailable for 4 of the 161 participants in the EFF set.
Measure: Number (95% Confidence Interval); unit: Percentage of regions
Groups:
- Central Reader 1: Central Reading Center 1
- Central Reader 2: Central Reading Center 2
- Central Reader 3: Central Reading Center 3
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of regions | 75.0 [62.10 to 84.60] | 68.9 [55.43 to 79.73] | 65.2 [53.40 to 75.38]

2. Primary Outcome: Patient-level Positive Predictive Value (PPV) (With Anatomical Localization) of Vidoflufolastat (18F)
Description: Patient-level positive predictive value (PPV) is defined as the percentage of participants who have at least one True Positive (TP) lesion (exactly localized correspondence between PET imaging and the reference standard), regardless of any co-existent False Positive (FP) findings, out of all participants who are PET/CT scan positive.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of participants | 76.5 [62.51 to 87.21] | 69.0 [55.46 to 80.46] | 64.6 [51.77 to 76.08]

3. Secondary Outcome: Patient-level Sensitivity of Vidoflufolastat (18F)
Description: Patient-level sensitivity is defined as the percentage of participants who test positive on vidoflufolastat (18F) and Composite Truth Standard (CTS) (True Positive (TP)) among those that are CTS positive (True Positive (TP) or False Negative (FN)).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of participants | 63.9 [50.63 to 75.84] | 66.7 [53.31 to 78.31] | 71.2 [57.92 to 82.24]

4. Secondary Outcome: Patient-level Specificity of Vidoflufolastat (18F)
Description: Patient-level specificity is defined as the percentage of participants who test negative on vidoflufolastat (18F) and CTS (True Negative (TN)) among those that are CTS negative (True Negative (TN) or False Positive (FP)).
Time Frame: as for outcome 1
Population: The Efficacy Analysis Set (EFF) included all enrolled participants who received the dose of investigational treatment (i.e. vidoflufolastat (18F)), had both an evaluable vidoflufolastat (18F) PET/CT scan and at least one evaluable CTS assessment, and did not receive any prohibited systemic antineoplastic therapy before the completion of PET/CT and surgery. Baseline PSA levels were unavailable for 4 of the 161 participants in the EFF set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of participants | 88.0 [79.98 to 93.64] | 82.2 [73.30 to 89.08] | 77.5 [68.11 to 85.14]

5. Secondary Outcome: Patient-level Negative Predictive Value (NPV) of Vidoflufolastat (18F)
Description: Patient-level negative predictive value is defined as the percentage of participants who are both vidoflufolastat (18F) and CTS negative (True Negative (TN)) among those who test negative on vidoflufolastat (18F) (True Negative (TN) or False Negative (FN)).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of participants | 80.0 [71.30 to 87.02] | 80.6 [71.62 to 87.72] | 82.3 [73.17 to 89.33]

6. Secondary Outcome: Patient-level Accuracy of Vidoflufolastat (18F)
Description: Patient-level accuracy is defined as the percentage of participants who are CTS and vidoflufolastat (18F) positive (True Positive (TP)) and negative (True Negative (TN)) among those participants that identified on vidoflufolastat (18F) (True Positive (TP), True Negative (TN), False Positive (FP) or False Negative (FN)).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of participants | 78.9 [71.76 to 84.91] | 76.4 [69.07 to 82.72] | 75.2 [67.74 to 81.62]

7. Secondary Outcome: Patient-level Correct Detection Rate (CDR)
Description: Patient-level correct detection rate (CDR) is defined as the percentage of participants who have at least one True Positive (TP) lesion (exactly localized correspondence between PET imaging and the reference standard), regardless of any co-existent False Positive (FP) findings, out of all participants who are scanned.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percenage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percenage of participants | 24.2 [17.83 to 31.59] | 24.8 [18.38 to 32.26] | 26.1 [19.49 to 33.58]

8. Secondary Outcome: Patient-level Detection Rate
Description: Patient-level detection rate is defined as the percentage of participants who have at least one PET positive lesion, regardless of True Positive (TP) or False Positive (FP) findings, out of all participants who are scanned.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of participants | 31.7 [24.58 to 39.46] | 36.0 [28.62 to 43.95] | 40.4 [32.72 to 48.38]

9. Secondary Outcome: Region-level Sensitivity of Vidoflufolastat (18F) (Overall)
Description: Region level sensitivity is defined as the percentage of regions that test positive on both vidoflufolastat (18F) and CTS (True Positive (TP)) among those regions that are CTS positive (True Positive (TP) or False Negative (FN)).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of regions
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of regions | 53.2 [42.19 to 63.85] | 58.2 [46.69 to 68.81] | 58.0 [47.07 to 68.25]

10. Secondary Outcome: Region Level Specificity of Vidoflufolastat (18F)
Description: Region level specificity is defined as the percentage of regions that test negative on both vidoflufolastat (18F) and CTS (True Negative (TN)) among those regions that are CTS negative (False Positive (FP) or True Negative (TN)).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of regions
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of regions | 98.1 [96.77 to 98.85] | 97.1 [95.61 to 98.16] | 96.5 [94.94 to 97.66]

11. Secondary Outcome: Region Level Negative Predictive Value (NPV) of Vidoflufolastat (18F)
Description: Region level negative predictive value is defined as the percentage of regions that are CTS and vidoflufolastat (18F) negative (True Negative (TN)) among those regions that test negative on vidoflufolastat (18F) (True Negative (TN) or False Negative (FN)).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of regions
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of regions | 95.1 [93.26 to 96.40] | 95.5 [93.76 to 96.82] | 95.4 [93.56 to 96.73]

12. Secondary Outcome: Region Level Accuracy of Vidoflufolastat (18F)
Description: Region level accuracy is defined as the percentage of regions that are CTS andvidoflufolastat (18F) positive (True Positive (TP)) and negative (True Negative (TN)) among those regions that identified on vidoflufolastat (18F) (True Positive (TP), True Negative (TN), False Positive (FP) and False Negative (FN)).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of regions
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 161 | 161 | 161
Percentage of regions | 93.7 [91.76 to 95.15] | 93.3 [91.32 to 94.86] | 92.7 [90.65 to 94.28]

13. Secondary Outcome: Patient-level Positive Predictive Value (PPV) of Vidoflufolastat (18F) Related to PSA Levels
Description: Patient-level positive predictive value related to PSA levels is defined as the percentage of participants who have at least one True Positive (TP) lesion (exactly anatomically localized correspondence between vidoflufolastat (18F) PET imaging and the reference standard), regardless of any co-existent False Positive (FP) findings, out of all participants who are vidoflufolastat (18F) positive, stratified by PSA levels. This endpoint was analyzed in each of the following subgroups: PSA ≤ 0.5 ng/mL; 0.5 ng/mL<PSA≤1 ng/mL; 1 ng/mL<PSA≤2 ng/mL; 2 ng/mL<PSA≤5 ng/mL; PSA > 5 ng/mL.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 157 | 157 | 157
Percentage of Participants
  Subgroup: PSA <= 0.5 ng/mL (n = 100,100,100): number analyzed (Participants) | 100 | 100 | 100
  Subgroup: PSA <= 0.5 ng/mL (n = 100,100,100) | 60.9 [38.54 to 80.29] | 59.3 [38.80 to 77.61] | 53.3 [34.33 to 71.66]
  Subgroup: 0.5 ng/mL <PSA <= 1 ng/mL (n = 29, 29, 29): number analyzed (Participants) | 29 | 29 | 29
  Subgroup: 0.5 ng/mL <PSA <= 1 ng/mL (n = 29, 29, 29) | 100 [66.37 to 100] | 66.7 [34.89 to 90.08] | 76.9 [46.19 to 94.96]
  Subgroup: 1 ng/mL <PSA <= 2 ng/mL (n = 11, 11, 11): number analyzed (Participants) | 11 | 11 | 11
  Subgroup: 1 ng/mL <PSA <= 2 ng/mL (n = 11, 11, 11) | 75.0 [34.91 to 96.81] | 71.4 [29.04 to 96.33] | 71.4 [29.04 to 96.33]
  Subgroup: 2 ng/mL <PSA <= 5 ng/mL (n=11,11,11): number analyzed (Participants) | 11 | 11 | 11
  Subgroup: 2 ng/mL <PSA <= 5 ng/mL (n=11,11,11) | 100 [54.07 to 100] | 100 [54.07 to 100] | 66.7 [29.93 to 92.51]
  Subgroup: PSA > 5 ng/mL (n = 6,6,6): number analyzed (Participants) | 6 | 6 | 6
  Subgroup: PSA > 5 ng/mL (n = 6,6,6) | 100 [39.76 to 100] | 100 [39.76 to 100] | 100 [39.76 to 100]

14. Secondary Outcome: Overview of Adverse Events (AEs) and Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
Time Frame: From first dosing (Day 1) up to 14 days post dosing
Population: Safety set (SAF): All participants who received at least one dose of vidoflufolastat (18F) or Gallium (68Ga) gozetotide.
  The vidoflufolastat (18F) Safety Set (F-SAF) included all participants who received the investigational treatment (i.e. vidoflufolastat (18F)).
  The gallium (68Ga) gozetotide safety Set (Ga-SAF) included all participants who received Gallium (68Ga) gozetotide.
Measure: Count of Participants; unit: Participants
Groups:
- Vidoflufolastat (18F): Participants received vidoflufolastat (18F) on Day 1 or Day 15 (investigational imaging agent of interest)
- Gallium (68Ga) Gozetotide: Participants received gallium (68Ga) gozetotide (as part of CTS if required, and for secondary endpoint) on Day 1 or Day 15
Arm/Group | Vidoflufolastat (18F) | Gallium (68Ga) Gozetotide
Number analyzed (Participants) | 171 | 178
Participants
  Adverse Events (AEs) | 20 | 16
  Treatment-related AEs | 6 | 2
  Serious Adverse Events (SAEs) | 1 | 0
  Treatment-related SAEs | 0 | 0
  Fatal serious AEs | 0 | 0
  Treatment-related fatal AEs | 0 | 0
  AEs leading to treatment discontinuation | 0 | 0
  Treatment-related AEs leading to treatment discontinuation | 0 | 0
  AEs leading to dose adjustment / interruption | 0 | 0
  AEs requiring additional therapy | 2 | 4

15. Secondary Outcome: Vidoflufolastat (18F) Scan Inter-reader Variability
Description: Inter-reader variability is defined as the agreement among three readers determination of vidoflufolastat (18F) images.
Time Frame: as for outcome 1
Population: The vidoflufolastat (18F) Safety Set (F-SAF) included all participants who received the investigational treatment (i.e. vidoflufolastat (18F)).
Measure: Number (95% Confidence Interval); unit: % agreement
Arm/Group | Vidoflufolastat (18F)
Number analyzed (Participants) | 171
% agreement | 65.5 [56.84 to 74.15]

16. Secondary Outcome: Vidoflufolastat (18F) Scan Intra-reader Variability
Description: Intra-reader variability is defined as the within-reader agreement for two different time points of vidoflufolastat (18F) images.
Time Frame: as for outcome 1
Population: The vidoflufolastat (18F) Safety Set (F-SAF) included all participants who received the investigational treatment (i.e. vidoflufolastat (18F)). Scans for a subset of 19 participants from the vidoflufolastat (18F) safety set were read by each reader at 2 different time points
Measure: Number (95% Confidence Interval); unit: % agreement
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 19 | 19 | 19
% agreement | 61.2 [10.39 to 100] | 100 [100 to 100] | 100 [100 to 100]

17. Secondary Outcome: Concordance Between Vidoflufolastat (18F) and Gallium (68Ga) Gozetotide for Detection of Lesions at Lesion Level Using Central Reads (Overall)
Description: Concordance between vidoflufolastat (18F) and gallium (68Ga) gozetotide for detection of PSMA-positive lesions (location and number) using central reads.
Time Frame: as for outcome 1
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of lesions
Groups:
- Central Reader 1: Central Reding Center 1
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 171 | 171 | 171
Percentage of lesions | 51.1 [40.62 to 61.49] | 48.2 [38.86 to 57.66] | 55.1 [44.41 to 65.36]

18. Secondary Outcome: Change in Patient Management Plans Attributed to the Vidoflufolastat (18F) PET/CT Scan
Description: Change in patient management plans attributed to the PET/CT scan is defined as the percentage of participants who underwent a change in intended treatment plan attributed to the vidoflufolastat (18F) PET/CT scan as assessed by pre and post imaging questionnaires.
Time Frame: From randomization up to 14 days after obtaining the results of the vidoflufolastat (18F) PET imaging
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Vidoflufolastat (18F)
Number analyzed (Participants) | 171
Participants | 61

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dosing (Day 1) up to 14 days post dosing.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up.
Arm/Group | Vidoflufolastat (18F) | Gallium (68Ga) Gozetotide
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/178
Serious Adverse Events (participants affected / at risk) | 1/171 | 0/178
Other Adverse Events (participants affected / at risk) | 20/171 | 16/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vidoflufolastat (18F) (N=171) | Gallium (68Ga) Gozetotide (N=178)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vidoflufolastat (18F) (N=171) | Gallium (68Ga) Gozetotide (N=178)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 5 | 0
Fatigue (General disorders) | 1 | 0
Injection site warmth (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Amylase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Apathy (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The participant cohort was mainly European and White, with only one site initiated in the USA. Furthermore, low participant numbers in some subgroups (i.e. participants with prior curative radiation therapy (RT) and participants with baseline Prostate-specific antigen (PSA) levels >1 ng/mL) precluded interpretation of subgroup analyses. In addition, Composite Truth Standard (CTS) Level 1 (histopathology) was only usable from a very small proportion of patients in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT04838613/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT04838613/SAP_001.pdf